CLINICAL TRIAL: NCT04817384
Title: Comparison of Immediate Effects of Graston Technique and Classical Massage in Primary School Children With Chronic Neck Pain
Brief Title: Graston Technique and Classical Massage for Chronic Neck Pain of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2020-0238
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Neck; Pain
Keywords: graston; massage; children; musculoskeletal
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston technique group (Experimental): For Graston practice, instruments made of stainless steel material of a type suitable for the body structures and sizes of the children will be preferred. The treatment time takes approximately 20-25 minutes depending on the area being treated. The instant effects of the people will be looked at.
  Interventions: Other: Classical Massage
- Classical massage group (Experimental): The trapezius, erector spina and levator scapula muscles will be applied with one hand or both hands, starting with general stroking. The intermediate to be used is baby oil or natural oils. The application time will be approximately 20 minutes.
  Interventions: Other: Graston technique

INTERVENTIONS:
Other: Graston technique — For Graston practice, children will be asked to sit with a support forward. Vaseline will be used as an intermediate during the application. Instruments made of stainless steel material of a type suitable for the body structures and sizes of the children will be preferred. Larger instruments will be used for larger areas and smaller for smaller regions and fibrocytic areas. The frequency of the plastering and friction movements will be applied in 60 repetitions per minute. While the graston technique is applied to individuals; Superficial muscles in the entire dorsal region will be included in the treatment. These muscles, respectively, the levator scapula, trapezius, and erroctor spina muscles were selected. The treatment time takes approximately 20-25 minutes depending on the area being treated. The instant effects of the people will be looked at.
  Arms: Classical massage group
Other: Classical Massage — In the neck massage application, the patient should be prepared, and the clothes in the upper back and neck area should be removed. The position of the patient will be in a sitting position with a pillow in front of him. The trapezius, erector spina and levator scapula muscles will be applied with one hand or both hands, starting with general stroking. The intermediate to be used is baby oil or natural oils. The application time will be approximately 20 minutes.
  Arms: Graston technique group

SUMMARY:
In reviews about manual therapy in children, mild, low-speed spinal mobilizations are emphasized as a safe treatment technique in infants, children and adolescents and have been used in clinics for years. Practices such as manipulation and manual therapy should adjust the force and speed used by the specialist practitioner in accordance with the age and developmental level of the child. Studies have emphasized that massage is an effective method in the treatment of chronic pain for children and adolescents. Significantly low pain and positive mood have been reported by children after these manual therapy sessions. Accordingly, the aim of the planned study is to compare the effects of graston technique and classical massage in children with chronic neck pain.

DETAILED DESCRIPTION:
Although there are new physiotherapy interventions for musculoskeletal pain, it is seen that studies about manual techniques are limited in childhood. Graston technique includes a small metallic instrument known as "strigil" and used for therapeutic purposes in ancient Greece and Rome. Another source is based on the traditional Chinese treatment known as "gua sha". Those who found the Graston technique are Dr. Konin, Dr. Greenstein, and Dr. Schrader. The basis of the Graston technique used today was inspired by James Cyriax. When the effects of the Graston technique are investigated, they aim to reduce pain, evaluate and increase soft tissue mobility, and improve range of motion and function. This technique is applied using specially designed curved stainless steel tools. These devices create micro trauma to restore normal elasticity and function in soft tissue. The different structures of the instruments allow to modify the degree of treatment. Small size instruments can be used on smaller anatomical structures and mild symptoms. Larger sized instruments are suitable for large treatment areas and severe conditions. Instruments are applied to the soft tissue at 30-60 degree angles with multi-directional stroking movements. The application time is applied for a maximum of 30 to 60 seconds per tissue site. In addition, whether the problem is acute or chronic is the most important factor that determines the duration of treatment. Total treatment time with instruments is generally minimum 8 minutes. It is applied with a maximum of 20 minutes.

In reviews about manual therapy in children, mild, low-speed spinal mobilizations are emphasized as a safe treatment technique in infants, children and adolescents and have been used in clinics for years. Practices such as manipulation and manual therapy should adjust the force and speed used by the specialist practitioner in accordance with the age and developmental level of the child. Studies have emphasized that massage is an effective method in the treatment of chronic pain for children and adolescents. Significantly low pain and positive mood have been reported by children after these manual therapy sessions. Accordingly, the aim of the planned study is to compare the effects of graston technique and classical massage in children with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* The children who have a chronic neck pain diagnosed by physician.
* The children who have minimum 10 degree limitation in at least one of neck movements.
* The children who have pain in neck region higher than 3 from Wong Baker pain scale.
* The children who state that they have neck pain for at least 3 months

Exclusion Criteria:

* The children who have other pain related to neurological or other orthopedic problem apart from neck region.
* The children who have any chronic disease requiring use of medicine like Hypertension and Diabetes Mellitus.
* The children who have open wound in neck region which may affect the interventions.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Level of Pain measured by Wong-Baker Faces Pain Rating Scale | change from baseline to immediately after the intervention
  The Wong-Baker Faces Pain Rating Scale is a pain scale that was developed by Donna Wong and Connie Baker. The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". The child will be asked to determine their level of pain according to this scale before and after the intervention.

SECONDARY OUTCOMES:
Pain Threshold measured by Pressure Algometry | change from baseline to immediately after the intervention
  Pressure algometry will be used to measure threshold. The pressure on the painful region is recorded in number (P).
Range of motions of neck joint measured by universal goniometer | change from baseline to immediately after the intervention
  Universal goniometer will be used for neck joint. Flexion, extension, lateral flexion and rotations will be recorded in degrees.
Satisfaction level from the application measured by VAS | immediately after the intervention
  The child will be asked to specify his/her satisfaction from the manual therapy (graston or classical massage) after the practice. The Visual Analogue Scale will be used to show the level. Zero will ne no any satisfaction and Ten will be too much satisfaction. The line starting from zere to ten cm will be given to child and asked to sign how much he/she is satisfied from the intervention.